CLINICAL TRIAL: NCT01112826
Title: Phase III Study of Adjuvant Capecitabine Metronomic Chemotherapy in Triple-negative Operable Breast Cancer
Brief Title: Efficacy of Capecitabine Metronomic Chemotherapy to Triple-negative Breast Cancer
Acronym: SYSUCC-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-001
Record Dates: First submitted 2010-04-22; First posted 2010-04-28 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer; metronomic chemotherapy; capecitabine (xeloda)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine (Experimental): Capecitabine 650 mg/m2 bid
  Interventions: Drug: Capecitabine
- Standard treatment (No Intervention): Treatment according to National Comprehensive Cancer Network (NCCN) guideline.

INTERVENTIONS:
Drug: Capecitabine — capecitabine 650 mg/m2 twice every day for 1 year.
  Arms: Capecitabine

SUMMARY:
The primary objective of this study is to compare disease-free survival (DFS) of patients with triple negative breast cancer randomised to treatment with standard adjuvant chemotherapy alone or to standard adjuvant chemotherapy followed by 1 year of Capecitabine (Xeloda) metronomic therapy.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) is an aggressive disease without tumor-specific treatment options. Patients with triple-negative disease had an increased likelihood of distant recurrence and death within 5 years of diagnosis. Median time to distant recurrence was significantly shorter. This study will evaluate the efficacy and safety of the addition of Capecitabine to standard adjuvant therapy in patients with triple negative breast cancer. Patients will be randomized to receive either standard chemotherapy (according to NCCN guideline), or standard chemotherapy followed by 1 year of metronomic Capecitabine (650mg/m2, twice every day). The anticipated time on study treatment is 12 months, and the target sample size is 432 individuals.Disease-free Survival (DFS) will be primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >=18 years of age;
* The patients must be Operable primary invasive breast cancer;
* Definitive loco-regional surgery must be completed;
* Primary tumor centrally confirmed as triple negative;
* Operable node-positive (or node-negative with tumor diameter ≥ 0.5cm);
* Chest, abdominal, bone imaging performed with 3 months prior to randomization must not reveal the presence of distant spread;
* There are normal organ function, including bone marrow function, renal function, liver function, and cardiac function;
* All patients must have signed and dated an informed consent form.

Exclusion Criteria:

* Patients with bilateral breast cancer, inflammatory carcinomas;
* Patients with positive supraclavicular or internal mammary lymph node;
* Previous breast cancer history;
* Any previous malignancy exceptions for carcinoma of the cervix, squamous carcinoma of the skin, or basal cell carcinoma of the skin;
* Pregnant or breast-feeding women;
* Women who are unwilling to agree to use an effective non-hormonal method of contraception during the treatment period of Xeloda;
* Any sex hormonal therapy;
* Malabsorption syndrome.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2010-04-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 36 months
  The final analysis are expected to occur 36 months after the end of recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Zhong-yu, MD, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan J, Bi XW, Hua X, Huang H, Cai L, Zhao L, Chen QJ, Chen XX, Wang XL, Lin Y, Zhang AQ, Zhong YY, Xu F, Huang JJ, An X, Shi YX, Wang X, Wang SS, Xue C, Yuan ZY. Metronomic capecitabine as extended adjuvant chemotherapy for early triple-negative breast cancer (SYSUCC-001): updated 10-year outcomes and post-hoc exploratory biomarker analysis from a randomised, phase 3 trial. Lancet Oncol. 2025 Dec;26(12):1575-1583. doi: 10.1016/S1470-2045(25)00545-5. PMID 41308674
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Wang X, Wang SS, Huang H, Cai L, Zhao L, Peng RJ, Lin Y, Tang J, Zeng J, Zhang LH, Ke YL, Wang XM, Liu XM, Chen QJ, Zhang AQ, Xu F, Bi XW, Huang JJ, Li JB, Pang DM, Xue C, Shi YX, He ZY, Lin HX, An X, Xia W, Cao Y, Guo Y, Su YH, Hua X, Wang XY, Hong RX, Jiang KK, Song CG, Huang ZZ, Shi W, Zhong YY, Yuan ZY; South China Breast Cancer Group (SCBCG). Effect of Capecitabine Maintenance Therapy Using Lower Dosage and Higher Frequency vs Observation on Disease-Free Survival Among Patients With Early-Stage Triple-Negative Breast Cancer Who Had Received Standard Treatment: The SYSUCC-001 Randomized Clinical Trial. JAMA. 2021 Jan 5;325(1):50-58. doi: 10.1001/jama.2020.23370. PMID 33300950